CLINICAL TRIAL: NCT01636063
Title: Mifepristone Versus Misoprostol for Cervical Preparation Prior to Surgical Abortion Between 11 to 15 Weeks
Acronym: MIMI11-15
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor subject enrollment
Sponsor: Boston University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SFPRF12-16
Record Dates: First submitted 2012-07-03; First posted 2012-07-10 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Induced Abortion; Abortion Techniques; Mifepristone; Misoprostol
Keywords: Induced Abortion; Abortion Techniques; Mifepristone; Misoprostol; Initial Cervical Dilation
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mifepristone (Experimental): Subjects will receive 200 mg of capsulized mifepristone orally for the purpose of cervical preparation before surgical abortion
  Interventions: Drug: Mifepristone
- Misoprostol (Active Comparator): Subjects will receive 400 mcg of buccal misoprostol for the purposes of cervical preparation.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — Mifepristone 200 mg capsulized orally once 24-48 hours prior to abortion procedure
  Other Names: RU-486
  Arms: Mifepristone
Drug: Misoprostol — Misoprostol 400 mcg buccally once 3 hours prior to abortion procedure
  Other Names: Cytotec
  Arms: Misoprostol

SUMMARY:
Surgical abortion in the late first trimester and early second trimester is usually performed with the aid of a cervical preparing agent, which helps to open up the uterine cervix for the procedure. Routine use of cervical preparants is recommended by several organizations during this period of pregnancy before surgical abortion, especially in younger women or those who have not delivered a baby, because their cervices may be more difficult to dilate without a preparant.

The standard medication used for cervical preparation is misoprostol. Unfortunately, misoprostol may cause uncomfortable uterine cramping and vaginal bleeding in patients who use it. Another medication called mifepristone has been shown to dilate the cervix better than misoprostol in the first trimester, but little information exists about using mifepristone in the late first trimester and early second trimester.

The investigators plan to perform a prospective, double-blind, randomized trial to evaluate if mifepristone is a better cervical preparant than misoprostol. A total of 110 participants who are pregnant women desiring pregnancy termination 11 to 15 weeks gestational age will be recruited. Half will receive mifepristone and the other half misoprostol. The investigators will measure the amount of cervical dilation achieved right before a surgical abortion to determine if mifepristone is significantly different than misoprostol as a cervical preparant at this stage of pregnancy. The investigators expect that mifepristone will work better than misoprostol for this purpose.

The investigators hope to generate information about mifepristone so that women and their health care providers can know more about mifepristone as an option for cervical preparation before surgical abortion.

DETAILED DESCRIPTION:
This study will use a prospective, double-blind, randomized clinical trial design. As our main objective is to determine whether one pharmacological method of cervical preparation is more effective than the other in our population, this is the most appropriate study design. A double-blinded, randomized trial will allow for the maximal prevention of bias affecting study results. The study will be structured as a two-tailed comparison, as it is possible that mifepristone is significantly less effective than misoprostol in effecting initial cervical dilation. While previous studies have indicated that mifepristone is superior to misoprostol in this regard, our study focuses on a later gestational age range. Therefore, we believe that a one-tailed comparison would be inappropriate to test whether there is a difference between mifepristone and misoprostol as cervical preparing agents in our gestational age range.

We will enroll approximately 50 subjects between 11 0/7 and 15 0/7 weeks GA seeking abortion and randomize them into two groups in a 1:1 ratio. Group A subjects will receive mifepristone 200 mg capsulized orally at the time of their preoperative visit and be given two folic acid tablets (misoprostol placebo) to place buccally on the day of their procedure. Group B subjects will receive empty capsules (mifepristone placebo) orally at the time of their preoperative visit and be given two misoprostol 200 mcg tablets to place buccally on the day of their procedure.

To preserve blinding, we will place mifepristone in capsules provided by the BMC IDS. Subjects not receiving mifepristone will receive identically-appearing empty capsules.

The study will take place at Boston Medical Center's outpatient Women's Care Center. Preoperative appointments will take place in the Pre-Procedure Unit (PPU) and abortion appointments will take place in the Gynecology Procedures Unit (GPU). Patients seeking abortion services at BMC will constitute the population that will be the source of the study sample. Because we seek to investigate mifepristone and misoprostol as cervical preparants in the population of women seeking abortion services, this is an appropriate population from which to sample.

Patients who are eligible to enroll as subjects in the investigation will be identified by the clinical provider who sees them for their preoperative visit. Approximately 20 patients per month seen at our clinic meet the criteria for inclusion into the study. The provider will describe the study briefly to the potential subject, and if they are interested, the provider will contact study staff. The staff member will describe the study in greater detail and obtain informed consent to take part in the study.

Subject allocation to treatment group will be double-blind. The Boston Medical Center Investigational Drug Service (IDS) will prepackage all study medications in a random order and sequentially number the packages.

We will enroll approximately 110 subjects between 11 0/7 and 15 0/7 weeks GA seeking abortion and allocate them randomly into two equal groups of subjects. Group A subjects will receive capsules containing mifepristone 200 mg orally at the time of their preoperative visit and be given two folic acid tablets (misoprostol placebo) to place buccally on the day of their procedure. Group B subjects will receive a empty capsules (mifepristone placebo) orally at the time of their preoperative visit and be given two misoprostol 200 mcg tablets to place buccally on the day of their procedure.

It is important to note that the investigation will use cervical preparants in a similar fashion to what is already standard practice at BMC. Mifepristone ingestion is directly observed by a clinic provider, while misoprostol is dispensed at the preoperative visit for the patient to place buccally herself approximately 3 hours before their abortion procedure. Patients between 11 and 12 weeks GA receive 400 mcg misoprostol buccally three hours prior to their procedure or no preparant, at the discretion of the surgeon. For patients between 12 and 14 weeks GA, 400 mcg buccal misoprostol for three hours prior to their procedure is the standard preparant. Patients between 14 and 15 weeks GA have the aforementioned misoprostol dosing option, and can instead also elect to receive mifepristone 200 mg orally 24 to 36 hours before their abortion procedure. Patients between 14 and 15 weeks GA can also elect to receive osmotic dilators as the cervical preparant method. Therefore, both agents used in our study are familiar to our clinicians and are already in use for patients at our facility in a similar fashion.

Enrolled subjects will be given a study subject number that corresponds to a treatment group assignment, which will be determined in advance by the BMC IDS in a random fashion. The clinic provider and study staff member will be blinded to the assignment, as will the subject. While the study is being conducted, only the BMC IDS will have access to the study subject treatment assignments. The clinic provider and study staff will then observe the subject take the first study agent (mifepristone or placebo). In order to preserve blinding, the BMC IDS will provide indistinguishable capsules of mifepristone and empty capsules.

They will then direct the patient to place the second study agent (misoprostol or placebo) buccally approximately three hours before their abortion procedure. This time will correspond to 6 am for morning procedures and 10 am for afternoon procedures. To preserve provider blinding, the second study agent will be in an opaque package. The BMC IDS is unable to provide indistinguishable versions of misoprostol and folic acid because we plan buccal use. Despite this, we do not anticipate a significant threat to subject blinding.

In order to ensure abortion provider blinding, the clinic provider and study staff member who enroll a subject will not be eligible to perform the subject's abortion.

At the subject's preoperative visit, the following data will be collected: Study subject number; date; age; race/ethnicity; ultrasound-confirmed gestational age; gravidity; parity; time of first study agent ingestion; history of prior live births; history of prior pregnancy loss; history of prior elective abortion; history of cervical dysplasia treatment procedures (cold knife cone, LEEP, cryotherapy).

A checklist of the aforementioned exclusion criteria will be present on the preoperative data sheet to prevent enrollment of subjects who meet these criteria.

One follow-up visit will be planned for all subjects: their abortion procedure appointment, which will occur 24 to 48 hours after their ingestion of the first study agent. At this encounter, all of the outcome variables will be measured and collected for data analysis. Once the subject arrives to the GPU, a study staff member will confirm and record the time of buccal placement of the second study agent. The subject will then undergo the routine intake process of all abortion patients in the GPU, which includes a preoperative safety screening by a registered nurse. After the intake process, the patient will undergo their abortion procedure no sooner than three hours after the buccal placement of the second study agent. For procedural anesthesia and analgesia, patients receiving care in the GPU have two choices. They may choose to receive IV conscious sedation, consisting of midazolam and fentanyl in addition to lidocaine paracervical block. The alternative is IM ketorolac and lidocaine paracervical block. Study participants will be afforded the same choice as other abortion patients. The abortion will then be performed, including assessment of initial cervical dilation, which is described below. The subject will then remain in the GPU recovery area until she meets criteria for discharge, consistent with guidelines in place for all patients receiving care in the GPU.

To measure initial cervical dilation, Pratt mechanical dilators will be used. Starting with a 43F Pratt dilator, attempts will be made to pass sequentially smaller diameter dilators until a dilator passes without resistance. The size of the largest dilator to pass without resistance will be recorded as the initial cervical dilation value. Using dilators from largest to smallest will avoid causing dilation during measurement of initial cervical dilation. This method of measuring initial cervical dilation has been described in published studies, including by Goldberg, et al. (19) Physicians who perform abortions for patients within the study will be trained to conduct the measurement of initial cervical dilation in a standard fashion.

All abortions will be performed by attending OB-GYN physicians and family planning fellows to limit confounding due to provider inexperience on the part of residents and medical students.

The data to be collected will include the date and time of buccal placement of the second study agent; subject's experience of preoperative vaginal bleeding, nausea, vomiting or diarrhea; preoperative pain score; anesthesia/analgesia agents used and doses used; initial cervical dilation; the amount of additional dilation needed to perform the procedure; intraoperative pain score; duration of procedure (speculum in to speculum out time); postoperative pain score; patient satisfaction; and provider rating of difficulty of procedure. Complications, if any, of the procedure will also be noted.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 years
* Fluency in English or Spanish
* Intrauterine pregnancy between 11 0/7 and 15 0/7 on the day of the abortion procedure
* Desire for pregnancy termination
* Ability to return for abortion procedure 24-48 hours after the preoperative visit

Exclusion Criteria:

* Allergy or contraindication to study agents
* Requirement of general anesthesia to perform the abortion
* Diagnosis of missed abortion, spontaneous abortion, incomplete abortion, or threatened abortion at time of initial preoperative evaluation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primary Investigator, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mifepristone | Misoprostol
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone | Misoprostol | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 15 | 18 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 13 | 21
  White | 11 | 6 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Initial Cervical Dilation at the Time of Surgical Abortion
Description: Initial cervical dilation as measured in French units by a Pratt cervical dilator prior to surgical abortion. The dilation was measured in French units with each French unit being equivalent to 0.33 mm.
Time Frame: 24 to 48 hours after enrollment
Measure: Mean (Standard Deviation); unit: French units
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 21 | 21
French units | 30.8 (6.8) | 31.1 (6.1)

ADVERSE EVENTS:
Arm/Group | Mifepristone | Misoprostol
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No